CLINICAL TRIAL: NCT07015606
Title: The Comparative Study of Sciatic Vs Femoral Nerve Mobilization Along With Electrical Muscle Stimulation in Low Back Pain
Brief Title: Sciatic Vs Femoral Nerve Mobilization With Electrical Muscle Stimulation for Treatment of Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ShalmarIHS
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain
Keywords: Low Back Pain (LBP)
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sciatic nerve mobilization with Electrical Muscle Stimulation (Other): Each patient will receive therapeutic sessions over 2 weeks (3 sessions per week), with total of 6 sessions. The repetition of mobilization will be 10 times for 2 sets with 2 minutes rest in between the sets. Electrical Muscle Stimulation (EMS) device was applied at a pulse frequency of 100 Hz. Placement of 2 surface electrodes will be used for stimulation over a session period of 15 minutes.
  Interventions: Other: Sciatic nerve mobilization with EMS
- Femoral neural mobilization with Electrical Muscle Stimulation (Other): Each patient will receive therapeutic sessions over 2 weeks (3 sessions per week), with total of 6 sessions. The repetition of mobilization will be 10 times for 2 sets with 2 minutes rest in between the sets. Electrical Muscle Stimulation (EMS) device was applied at a pulse frequency of 100 Hz. Placement of 2 surface electrodes will be used for stimulation over a session period of 15 minutes.
  Interventions: Other: Femoral neural mobilization with EMS

INTERVENTIONS:
Other: Sciatic nerve mobilization with EMS — Patients in both groups will receive electrical muscle stimulation. In addition, the group A will receive sciatic neural mobilization and group B will receive femoral neural mobilization. Patients were not allowed to take medication for pain during the study or to receive any other form of treatment outside the study. EMS device was applied at a pulse frequency of 100 Hz. Placement of 2 surface electrodes will be used for stimulation over a session period of 15 minutes. The repetition of mobilization will be 10 times for 2 sets with 2 minutes rest in between the sets. The frequency of Electrical muscle stimulation and the duration of neural mobilization will be increased after every session up to 10 Hz and 3 mints respectively.
  Arms: Sciatic nerve mobilization with Electrical Muscle Stimulation
Other: Femoral neural mobilization with EMS — Patients in both groups will receive electrical muscle stimulation. In addition, the group A will receive sciatic neural mobilization and group B will receive femoral neural mobilization. Patients were not allowed to take medication for pain during the study or to receive any other form of treatment outside the study. EMS device was applied at a pulse frequency of 100 Hz. Placement of 2 surface electrodes will be used for stimulation over a session period of 15 minutes. The repetition of mobilization will be 10 times for 2 sets with 2 minutes rest in between the sets. The frequency of Electrical muscle stimulation and the duration of neural mobilization will be increased after every session up to 10 Hz and 3 mints respectively.
  Arms: Femoral neural mobilization with Electrical Muscle Stimulation

SUMMARY:
to determine the therapeutic effectiveness of sciatic nerve mobilization compared to femoral nerve mobilization along with electrical stimulation in promoting functional recovery and alleviating symptoms in patients with low back pain and to reveal which one is more effective for pain relief and functional improvement in low back pain patients.

DETAILED DESCRIPTION:
Low back pain is a multi-dimensional musculoskeletal condition resulting in discomfort and functional limitation, arising from lower lumbar region radiating towards posterior lower limb or anterior thigh, often resulting from numerous factors like mechanical, degenerative, neuropathic, inflammatory, infectious, neoplastic and psychological factors. One of the most prevalent association of low back pain is nerve irritation and poor neuromuscular coordination. According to nerve pathway and innervation pattern, the main constituents of lumbosacral plexus are sciatic and femoral nerves. Sciatic nerve arises from L4-S3 spinal nerve roots passing through the gluteal region and down the posterior thigh innervating hamstrings, gastrocnemius, soleus, tibialis posterior, flexor digitorum longus, flexor hallucis longus, fibularis longus and brevis. Whereas, femoral nerve originates from L2-L4 and supply along the anterior region of thigh musculature like quadriceps femoris, sartorius, pectineus.

Normal nerve function, reduced mechanical sensitivity, and relief of radiating symptoms are the main goals of neural mobilization. Complementary to this, there are numerous studies which shows the effects of Electrical Muscle Stimulation that reduces pain by maximizes neuromuscular control and activation, facilitates blood circulation and prevents muscular atrophy in low back pain patients.

According to study conducted in 2022 by Romero-Morales and colleagues in Spain, neural mobilization has great effect in management of pain and disability in musculoskeletal disorders. Another study done in Japan in 2023 has describe the efficacy of Neural Mobilization on Pain, Mobility, and Psychosocial Functioning of Patients.

Peripherally neural mobilization increases nerve conductivity and physiologically it changes central sensitization. With an eye towards maximizing functional recovery and pain relief, this comparative study evaluates the combined effects of nerve mobilization and Electrical Stimulation in treatment of Low Back Pain, which has emerging evidence from a study which is published in the journal of pain, USA in 2002 that explains the efficacy of Electrical stimulation with combined therapy .

Another number of studies has also been done explaining the effect of neural mobilization on low back pain one of which is published in Pakistan journal of medical and health sciences in 2022 concluding that sciatic nerve mobilization is an effective treatment for pain and disability in patients.

With a lifetime prevalence in around 80% of adults, low back pain affects approximately 7.5% of the world's population and is the most often reported cause of long term impairment. Recent studies reveal that in Pakistan, particularly among manual laborers, healthcare professionals, and office workers, prevalence of low back pain increases from 30% to 50%.

Poor ergonomics, limited access to rehabilitation and ignorance, all these factors contribute in escalating incidence rate in Pakistan. Evidence based physiotherapeutic interventions are required to reduce the socioeconomic impact of low back pain, which is emerging in importance and is frequently connected with muscular weakness and decreased neural mobility. One of the most commonly reported causes of impairment worldwide is Low back pain that targets the femoral and sciatic nerves, results from mechanical stress on the lumbar plexus.

Techniques of neural mobilization aim to relieve pain, inflammation and normalize nerve mechanics. In addition to being used, it promotes blood circulation, muscle function rehabilitation and supports recovery of neural function. Electrical muscle stimulation aids in both sciatic and femoral nerve mobilizations clinically and direct their therapeutic effect on Low Back Pain. Therapeutic results can be affected by the anatomical and physiological differences between the two nerves. Electrical stimulation and neural mobilization can promote neuromuscular rehabilitation by their synergistic advantages. Finding the best approach makes it possible to have more clinically relevant evidence based therapies for low back pain management. This study aims to provide the evidence based intervention for the effective treatment of low back pain in Pakistan by examining the effectiveness of electrical muscle stimulation alone with sciatic and femoral nerve mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-50 years
* Radiating pain pattern
* Muscular pain pattern
* Negative sensory and motor neural examination
* Patients with peripheral nerve sensitization were included if they were adults and had leg pain duration of < 3 months(8)
* VAS Score between 4 and 8
* Positive findings of tests like thigh thrust, Patrick's Faber test, Gaenslen's test, modified Trendelenburg's test and Slump test.

Exclusion Criteria:

* Pregnancy
* Post-partum females
* Serious spinal pathology
* Sensory and motor deficient
* History of back and lower extremity surgery
* Patients with contraindication to Electrical Stimulation
* Any serious kind of co-morbidities like malignancy, infections
* Any kind of disability

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-08-28 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-11-29 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 8 WEEKS
  Pain intensity was further measured using the Visual Analog Scale (VAS), ranging from 0 mm (no pain) to 100 mm (worst imaginable pain). VAS scores were categorized as follows: 0-4 mm indicating no pain, 5-44 mm mild pain, 45-74 mm moderate pain, and 75-100 mm severe pain.21

SECONDARY OUTCOMES:
Oswestry disability index (ODI) | 8 WEEKS
  The Oswestry Disability Index (ODI) is a 10-item, patient-reported questionnaire used to assess functional impairment from lower back pain in both acute and chronic conditions. Disability levels are categorized from minimal to crippling, with scores ranging from 0-100. Each item is scored from 0 to 5, yielding a total score with a cut of ≤50.
Goniometer for range of motion (ROM) | 8 WEEKS
  Using a goniometer is a standard clinical method to assess hip joint mobility through active (patient-driven) or passive (clinician-assisted) movement. Normal ranges include hip flexion (0°-120°), abduction (0°-45°), and extension (0°-30°). Values below 110° for flexion, 35° for abduction, or 20° for extension may indicate functional limitation
EuroQol 5 Dimension Questionnaire (EQ-5D) | 8 WEEKS
  The EQ-5D is a standardized questionnaire used to assess health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 3- or 5-level scale, generating a health state index. Scores typically range from -0.594 to 1, where 1 indicates full health and <0.5 suggests poor health status. It aids in clinical evaluation, economic analysis, and treatment outcomes.